CLINICAL TRIAL: NCT00527553
Title: The Effect of Modified Eggs and Egg Products on the Measurable Macular Pigment in Healthy Subjects
Brief Title: The Effect of Eggs and Egg Products on Macular Pigment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: SenterNovem (Unknown); Newtricious BV (Unknown); Globus Ei BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 061127
Record Dates: First submitted 2007-09-03; First posted 2007-09-11 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2008-11

CONDITIONS: Age-related Macular Degeneration
Keywords: Macular pigment; AMD; ARM
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): daily consumption of a regular egg
  Interventions: Dietary Supplement: not enriched egg
- B (Experimental): daily consumption of a lutein-enriched egg, eggs laid by chickens on a lutein-enriched feed.
  Interventions: Dietary Supplement: lutein
- C (Experimental): daily consumtion of a zeaxanthin-enriched egg, eggs laid by chickens on a zeaxantin-enriched feed.
  Interventions: Dietary Supplement: zeaxanthin
- D (Experimental): daily egg product from enriched eggs
  Interventions: Dietary Supplement: egg product from enriched eggs
- E (No Intervention): control subjects were not blinded as they did not receive any aditional supplementation. Only markers measured during the trial period as a control.

INTERVENTIONS:
Dietary Supplement: not enriched egg — daily consumption of a regular egg, not enriched with either lutien nor zeaxanthin
  Arms: A
Dietary Supplement: lutein — daily lutein enriched egg
  Arms: B
Dietary Supplement: zeaxanthin — daily zeaxanthin enriched egg
  Arms: C
Dietary Supplement: egg product from enriched eggs — daily egg product from lutein enriched eggs
  Arms: D

SUMMARY:
Age-related macula degeneration (AMD, encompassing both dry and wet form), the late stage of Age-related maculopathy (ARM), is the leading cause of blindness in many developed countries in older persons (usually over 60 years of age). Visual compromise rises exponentially after the age of 70 with a 5-year incidence of around 1%. Studies have shown a possible protective effect of lutein on progression of AMD, where visual acuity improves after increased lutein intake. The incidence of bilateral AMD in persons with unilateral late ARM observed over a period of 10 years is over 50% with a 2.1-2.8% overall incidence in the study population.

Blue light hazard (excitation peak 440 nm) was shown to have a major impact on photoreceptor and RPE function inducing photochemical damage and cellular apoptosis, leading to retinal degeneration in an animal study. The current belief is that lutein accumulated in the macular region helps in the prevention of blindness by absorbing blue light and protecting the retina from oxidative stress. With the lipid matrix of the egg yolk being a proven vehicle for the efficient absorption of dietary lutein, it might be possible to increase plasma levels of lutein to therapeutic levels and control or prevent AMD. This, the investigators hope, will be accomplished by means of filtering out harmful blue light and the scavenging of free radicals by lutein and zeaxanthin.

DETAILED DESCRIPTION:
This will be a randomized placebo-controlled trial. The total study time will be two years of which 3 months are actual trial and follow-up time. Every individual will have 3 measuring points at set intervals. At every measuring point (days 1, 45 and 90), these subjects will undergo 6 different non-invasive measuring techniques. These are the mean visual acuity test using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart, contrast sensitivity using the Pelli-Robson chart, Scanning Laser Ophthalmoscope (SLO), Optical Coherence Tomography (OCT) and Heterochromatic Flicker Photometry (HFP) and the Reflectometer. A questionnaire will be taken at the beginning of the trail. The invasive part of the study involves blood sampling at all three times, measuring the serum concentration of lutein, zeaxanthin, omega-3 and lipoprotein using the HPLC analysis.

ELIGIBILITY:
Inclusion Criteria:

* No history of ARM or AMD
* 18 years and older
* Non-smoker
* No ocular media opacity
* Uses no nutritional supplements containing Lutein, Zeaxanthin or Omega-3
* BMI < 30
* No known cardiovascular disease

Exclusion Criteria:

* Diabetes
* Other known eye disease
* Known lipid metabolism disease
* Blood lipid level modifiers (e.g., Statin)
* Known allergy to eggs or egg products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Measurable macular pigment | 3 months

SECONDARY OUTCOMES:
Plasma Lutein and zeaxanthin concentrations, lipid profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: T. T.J. Berendschot, Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hostpital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Kelly ER, Plat J, Haenen GR, Kijlstra A, Berendschot TT. The effect of modified eggs and an egg-yolk based beverage on serum lutein and zeaxanthin concentrations and macular pigment optical density: results from a randomized trial. PLoS One. 2014 Mar 27;9(3):e92659. doi: 10.1371/journal.pone.0092659. eCollection 2014. PMID 24675775